CLINICAL TRIAL: NCT06879873
Title: MRD-Guided Surveillance in Operable Colon Adenocarcinoma (I-III)
Brief Title: MRD-Guided Surveillance in Operable Colon Adenocarcinoma (I-III)(SURVEILLANCE-I)
Acronym: SURI
Status: Not yet recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xu jianmin, Director of Colorectal Surgery Department, Zhongshan hospital, Fudan University, Fudan University
Other Study IDs: SURVEILLANCE-I
Record Dates: First submitted 2025-03-11; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Colorectal Cancer (CRC)
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — In this study, the specific types of samples that will be retained are peripheral blood samples collected from patients at multiple time points. These samples will be used for circulating tumor DNA (ctDNA) analysis to assess minimal residual disease (MRD) status.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- MRD-Guided Surveillance of I-III CRC

SUMMARY:
This study aims to explore the relationship between minimal residual disease (MRD) status and disease recurrence in patients with stage I-III operable colon adenocarcinoma. MRD refers to the presence of cancer cells that remain in the body after treatment but are undetectable by traditional imaging methods. The study will use a blood-based test to detect circulating tumor DNA (ctDNA) and assess its ability to predict cancer recurrence and survival outcomes.

Patients who are newly diagnosed with stage I-III colon adenocarcinoma and are eligible for surgery will be enrolled. Blood samples will be collected at multiple time points, including before surgery, after surgery, and during follow-up visits over three years. The study will compare MRD status with recurrence-free survival (RFS), overall survival (OS), and the time it takes for MRD to detect recurrence compared to standard imaging methods.

The goal is to determine whether MRD monitoring can provide early warning of cancer recurrence and help guide treatment decisions. This study may offer valuable insights into improving postoperative surveillance and personalized treatment strategies for colon cancer patients.

DETAILED DESCRIPTION:
This is a multicenter, prospective, observational study designed to evaluate the effectiveness of ctDNA-based MRD monitoring in predicting disease recurrence and survival outcomes in patients with stage I-III operable colon adenocarcinoma. The study will enroll 390 patients who have not previously received chemotherapy, radiotherapy, or targeted therapy.

Key Objectives:

Primary Objective:

To explore the correlation between MRD status and recurrence-free survival (RFS) in stage I-III colon adenocarcinoma patients.

Secondary Objectives:

To assess the relationship between MRD status and 1-year/2-year recurrence-free survival (1yRFS, 2yRFS).

To evaluate the association between MRD status and overall survival (OS).

Exploratory Objective:

To determine the average time by which MRD detection precedes imaging-based detection of disease recurrence.

Study Design:

Patients will undergo blood sampling at baseline (pre-surgery), post-surgery (7±2 days), and during follow-up visits at 1, 3, 6, 9, 12, 18, 24, and 36 months.

MRD status will be assessed using ctDNA methylation-based PCR technology, which offers a rapid and cost-effective alternative to traditional NGS-based methods.

Statistical Analysis:

The study will use Kaplan-Meier survival analysis to estimate RFS and OS.

Cox regression models will be employed to determine whether MRD status can serve as a prognostic factor for disease recurrence.

Ethical Considerations:

The study adheres to the principles of the Declaration of Helsinki and Chinese Good Clinical Practice (GCP) guidelines.

Informed consent will be obtained from all participants, and their privacy and confidentiality will be strictly maintained.

Expected Outcomes:

The study aims to validate the clinical utility of ctDNA-based MRD monitoring in predicting recurrence and survival outcomes, potentially offering a more effective tool for postoperative surveillance and treatment planning in colon cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age range: 18-80 years old, male or female not limited;
2. Histologically confirmed colon adenocarcinoma (i.e. adenocarcinoma, including adenocarcinoma, mucinous adenocarcinoma, signet ring cell carcinoma, undifferentiated carcinoma; excluding adenosquamous cell carcinoma);
3. Preoperative staging of stages I-III, without undergoing endoscopic ESD or EMR surgical resection;
4. Not receiving chemotherapy, radiotherapy, targeted therapy, or other anti-tumor treatments;
5. Radical surgery can be performed;
6. ECOG score 0-1 points;
7. The subjects voluntarily joined this study and signed an informed consent form, demonstrating good compliance and actively cooperating to return to the hospital for regular clinical follow-up diagnosis and treatment.

Exclusion Criteria:

1. Previously suffered from other malignant tumors (including non adenocarcinoma colorectal cancer);
2. Pregnant and lactating women;
3. According to the researchers' assessment, the patient also suffers from other diseases that may affect follow-up and short-term survival
4. Subjects have other factors that may lead to the forced termination of this study, such as other serious diseases (including mental illness, infectious diseases, fever ≥ 38 ℃, etc.) requiring combined treatment, serious laboratory examination abnormalities, accompanied by family or social factors, which will affect the safety of subjects, or the collection of data and samples.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients diagnosed with stage I-III resectable colon adenocarcinoma who have not received prior treatment. Participants will be recruited from multiple clinical centers and must meet specific eligibility criteria to ensure the study's validity.
  Key Characteristics of the Study Population:
  Diagnosis: Histologically confirmed colon adenocarcinoma (including adenocarcinoma, mucinous adenocarcinoma, signet-ring cell carcinoma, and undifferentiated carcinoma; excluding adenosquamous carcinoma).
  Stage: Clinical stage I-III, confirmed by preoperative imaging and clinical assessment.
  Treatment History: No prior chemotherapy, radiotherapy, targeted therapy, or other anti-cancer treatments.
  Surgical Eligibility: Candidates must be eligible for curative-intent surgery. General Health Status: ECOG performance status 0-1, indicating good functional status.
  Age Range: 18 to 80 years old. Consent & Compliance: Participants must provide informed consent and be willing
Sampling Method: Non-Probability Sample
Enrollment: 390 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Exploring the correlation between MRD status and disease recurrence rate (RFS) in stage I-III operable colon adenocarcinoma | From surgery until disease recurrence or up to 36 months, whichever occurs first
  Exploring the correlation between MRD status and disease recurrence rate (RFS) in stage I-III operable colon adenocarcinoma

SECONDARY OUTCOMES:
The correlation between MRD status and 1-year recurrence free survival (1yRFS) | From surgery until 12 months post-surgery
  The correlation between MRD status and 1-year recurrence free survival (1yRFS)
The correlation between MRD status and 2-year recurrence free survival (2yRFS) | From surgery until 24 months post-surgery
  The correlation between MRD status and 2-year recurrence free survival (2yRFS)
The correlation between MRD status and overall survival (OS) | From surgery until death or up to 36 months, whichever occurs first
  The correlation between MRD status and overall survival (OS)

OTHER OUTCOMES:
MRD detects disease recurrence earlier than imaging (CT) on average | From surgery until disease recurrence or up to 36 months, whichever occurs first
  MRD detects disease recurrence earlier than imaging (CT) on average

IPD SHARING:
Plan to Share IPD: No